CLINICAL TRIAL: NCT02472067
Title: A Pilot Study to Test the Efficacy of Psychologically-Based Physical Therapy Training for Treating Deployed U.S. Sailors and Marines With Musculoskeletal Injuries
Brief Title: Psychologically-Based Physical Therapy Treatment for Deployed U.S. Sailors and Marines With Musculoskeletal Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-01166
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Musculoskeletal Injury
Keywords: Musculoskeletal Injury; physical therapy; psychological intervention; risk factors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy (No Intervention): Usual care of physical therapy and rehabilitation for a musculoskeletal injury. Patients complete self-rated standardized surveys before and following treatment.
- Psychologically-Based Physical Therapy (Experimental): Psychologically-Based Physical Therapy includes the early identification and management of psychological obstacles to recovery in order to modify maladaptive responses previously found to be associated with chronicity and disability. This is accomplished through patient education, an emphasis on functional goals and encouraging self-care techniques. Patients complete self-rated standardized surveys before and following treatment.
  Interventions: Behavioral: Psychologically - Based Physical Therapy

INTERVENTIONS:
Behavioral: Psychologically - Based Physical Therapy — Psychologically - Based Physical Therapy targeting risk factors for disability.
  Arms: Psychologically-Based Physical Therapy

SUMMARY:
The main objective of this pilot project is to demonstrate the effectiveness of a psychologically-based physical therapy (PBPT) intervention for the prevention of disability in Active Duty Service Members who sustained a musculoskeletal injury (MSI) during deployment in support of combat operations on a carrier. This intervention is intended to optimize recovery and restore function in injured Active Duty Service Members.

The three aims necessary to accomplish the main objective are:

1. Demonstrate the feasibility of implementing PBPT on board a carrier;
2. Document and compare risk factors related to disability from MSI aboard two carriers;
3. Demonstrate the effectiveness of the PBPT intervention in a comparative effectiveness trial

DETAILED DESCRIPTION:
Musculoskeletal injuries pose a significant problem for Active Duty Service Members and are the main reason for separation and long-term disability. Little information exists on the determinants of disability and seeking care patterns in Sailors and Marines who experience MSI during deployment in support of combat operations, despite the fact that these branches of the armed services have the highest level of attrition from these disorders of all branches PBPT implemented in this setting has the potential to have a dramatic impact on the study outcomes. It is expected that an intervention of psychologically-based physical therapy targeting the common psychological risk factors (yellow flags) that include fear of activity including work, psychological distress, and perceived disability will be effective in reducing these risk factors and optimizing recovery and restoring function in the intervention group. Active Duty Service Members who seek care for a MSI on a carrier will benefit from early care by a trained physical therapist, which will reduce the likelihood of the formation or maintenance of maladaptive beliefs about injury previously found to be associated with disability.

The proposed study design is a quasi-experimental, pre-post- test with a non-concurrent control group to test the effectiveness of psychologically-based physical therapy aboard a US Navy Aircraft Carrier.

This approach will consist of one deployed carrier serving as the intervention and a second carrier serving as a control. The two carriers (intervention and equivalent control) will be chosen based on deployment schedules. Both carriers will have similar deployment characteristics to include; length of deployment, crew size and deployed health care team. For the purposes of this project, measurements will be done during deployment (pre physical therapy intervention and one month after enrollment) and after deployment. Thus, two different endpoints will be used, a post treatment endpoint (one month after enrollment), and a second which takes place after the carrier returns from deployment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting to medical for a primary complaint of a new MSI. A new MSI is considered in this study when the subject has not sought treatment for a period of 30 days or more prior to presenting to medical.

Exclusion Criteria:

* Subjects not eligible include those who require medical evacuation, or have a trauma/ comorbidities that may prevent them from receiving physical therapy treatment (i.e. amputations, fractures, contusions and other 'Red Flags' that required specialized medical care).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Psychological Distress (STarT Back Generic Screening Tool) | Change from baseline to one month following treatment.
  Measured using the STarT Back Generic Screening Tool.
Expectations of Recovery (single item question ) | Change from baseline to one month following treatment.
  Measured using a single item question constructed by the research team.
Self-Efficacy (COMI) | Change from baseline to one month following treatment.
  Measured using adapted questions from the Core Outcome Measurements Index (COMI).
Fear Of Work Activity (STarT Back Screening Tool) | Change from baseline to one month following treatment.
  Measured using questions adapted from the STarT Back Screening Tool.
Quality of Life (SF-12) | Measured one month following treatment.
  Measured using questions adapted from Short Form Health Survey(SF-12)
Perceived Disability (COMI) | Change from baseline to one month following treatment.
  Measured using adapted questions from the Core Outcome Measurements Index (COMI).
Pain Interference (DVPRS) | Change from baseline to one month following treatment.
  Measured using the Defense and Veterans Pain rating Scale (DVPRS).
Satisfaction with Process of Care (MRPS) | Measured one month after treatment.
  Measured using the MedRisk Instrument for Measuring Patient Satisfaction (MRPS)
Outcome Satisfaction (COMI) | Measured one month after treatment.
  Measured using adapted questions from the Core Outcome Measurements Index (COMI).

SECONDARY OUTCOMES:
Health Care Utilization (AHLTA) | Measured at six month follow-up
  Measured using the Armed Forces Health Longitudinal Technology Application (AHLTA).
Limited Duty (MEDBOLTT Database) | Measured at six month follow-up
  Measured using the MEDBOLTT Database.

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Weiser-Horwitz, PhD, Principal Investigator — NYU Medical Centre and School of Medicine

REFERENCES:
- [Background] Campello M, Ziemke G, Hiebert R, Weiser S, Brinkmeyer M, Fox B, Dail J, Kerr S, Hinnant I, Nordin M. Implementation of a multidisciplinary program for active duty personnel seeking care for low back pain in a U.S. Navy Medical Center: a feasibility study. Mil Med. 2012 Sep;177(9):1075-80. doi: 10.7205/milmed-d-12-00118. PMID 23025138
- [Background] Ziemke GW, Campello M, Rennix CP, Keer S, Zook J, Nordin M, et al. Retrospective Administrative Limited Duty Outcome Review Lovelace Respiratory Research Institute; 2012. Report No.: Contract Number 2011.029
- [Background] Hiebert R, Campello MA, Weiser S, Ziemke GW, Fox BA, Nordin M. Predictors of short-term work-related disability among active duty US Navy personnel: a cohort study in patients with acute and subacute low back pain. Spine J. 2012 Sep;12(9):806-16. doi: 10.1016/j.spinee.2011.11.012. Epub 2012 Jan 9. PMID 22227177